CLINICAL TRIAL: NCT02859584
Title: ASSESSMENT OF ADRENAL FUNCTION IN PATIENTS WITH ACUTE HEPATITIS USING CONCENTRATION OF SERUM TOTAL CORTISOL, SERUM FREE AND SALIVARY CORTISOL
Brief Title: ADRENAL FUNCTION IN PATIENTS WITH ACUTE HEPATITIS
Acronym: CORT-HEPAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2011-A00385-36
Record Dates: First submitted 2016-07-28; First posted 2016-08-09 (Estimated); Last update posted 2016-08-19 (Estimated); Status verified 2016-07

CONDITIONS: Acute Hepatitis
Keywords: Acute hepatitis; acute liver failure; adrenal dysfunction; salivary cortisol; serum free cortisol
MeSH Terms: conditions — Liver Failure, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- no serious acute hepatitis (Other)
  Interventions: Biological: Measure OF SERUM TOTAL CORTISOL, SERUM FREE AND SALIVARY CORTISOL
- Serious acute hepatitis (Other)
  Interventions: Biological: Measure OF SERUM TOTAL CORTISOL, SERUM FREE AND SALIVARY CORTISOL
- Healthy volunteers (Other)
  Interventions: Biological: Measure OF SERUM TOTAL CORTISOL, SERUM FREE AND SALIVARY CORTISOL
- Surrenal insufficiency (Other)
  Interventions: Biological: Measure OF SERUM TOTAL CORTISOL, SERUM FREE AND SALIVARY CORTISOL

INTERVENTIONS:
Biological: Measure OF SERUM TOTAL CORTISOL, SERUM FREE AND SALIVARY CORTISOL

SUMMARY:
A high frequency of adrenal dysfunction (AD) has been reported in severe acute hepatitis (SAH) using the dosage of serum total cortisol (STC). Because 90% of circulating serum cortisol is bound to proteins that are altered in SAH, we aimed to investigate the effect of decreased cortisol-binding proteins on STC, serum free cortisol (SFC) and salivary cortisol (SalivCort) in SAH.

Baseline (T0) and cosyntropin-stimulated (T60) STC, SFC and SalivCort concentrations were measured

DETAILED DESCRIPTION:
We prospectively and consecutively enrolled 75 patients suffering from a SAH (n=44) or a NSAH (n=31). Inclusion criteria were patients aged between 18 and 75 years with an acute hepatitis defined by an abrupt rise in serum aminotransaminase levels during the 15 previous days (AST or ALT greater than 500 IU/L or greater than 10 times the upper normal value); the acute hepatitis was considered as severe if the prothrombin index was lower than 50% and as non-severe if it was greater than 50%. We excluded patients with the following conditions: a history of hypothalamic-pituitary or adrenal disease, corticosteroids treatment within the previous 6 months, ketoconazole intake, oral candida infection, any visible bleeding in the oral cavity, liver transplanted patients, acute alcoholic hepatitis and night workers. Twenty-nine healthy controls (HC) were thereafter enrolled and similarly distributed with the SAH group on age, sex and estrogen pill intake, estrogen therapy being the most common cause for changes in CBG levels. HC were without any known illnesses and were not receiving any medications. To evaluate the range of the SFC concentrations, eight patients with a known AD caused by impairment of hypothalamic-pituitary-adrenal axis (n=5) and adrenal gland (n=3) and followed at the Endocrinology Department of Besancon were also studied.

STC, SFC and salivary cortisol concentrations were measured blindly before (T0 between 8am and 9am) and 60 minutes after (T60) an intravenous injection of 250 µg tetracosactrin (synacthenÒ, Sigma-Tau laboratory, France). Serum CBG, albumin and ACTH were also measured

ELIGIBILITY:
Inclusion Criteria:

* Inclusion of 101 test subjects and for statistical analysis:

  * 29 patients with non-acute severe hepatitis (TP> 50% and AST or ALT> 500 IU / L or> 10 xN for less than 15 days).
  * 43 patients with severe acute hepatitis (TP <50%). Patients with suspected IS with the assay of the CTS will retested at Synacthène 4 to 6 months later (10 desired subjects).
  * 29 healthy volunteers (control group included in the analysis).
* Inclusion of 10 patients with established IS (control group to estimate the low values of cortisol).
* Patient who signed the consent of study participation

Exclusion Criteria:

* Women during pregnancy or breastfeeding
* Minor and over 75 years
* Major protected within the meaning of Huriet
* Subject healthy volunteers in a sport competition
* Patients transplanted, HIV infection (also refusing HIV status) or patients on immunosuppressive therapies (including corticosteroids)
* ketoconazole Shot, rifampicin, mifepristone, megestrol or etomidate
* Treatment with corticosteroids irrespective of the route of administration
* severe acute alcoholic hepatitis
* oral fungal infection
* upper gastrointestinal bleeding or oral bleeding (contamination salivettes)
* unbalanced Diabetes
* unbalanced Hypertension
* Chronic heart failure (stage III or IV of the classification of the New York Heart Association [NYHA])
* Inability to receive clear information in patients with severe encephalopathy and do not have someone you trust
* Refusal of the participation agreement by signing the form of information and consent as defined in the protocol.
* exclusion period from another biomedical study
* Septic shock

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2011-08; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Concentration of the serum total cortisol (STC) in SAH. | 2 years
Concentration of the serum free cortisol (SFC) in SAH. | 2 years
Concentration of the salivary cortisol (SalivCort) in SAH. | 2 years

REFERENCES:
- See also: article — http://www.ncbi.nlm.nih.gov/pubmed/21281437